CLINICAL TRIAL: NCT06797349
Title: Determination of the Postprandial Glycemic Response and Glycemic Index of Nutritional Products: A Randomized Controlled Clinical Trial in Healthy Individuals
Brief Title: Glin4: Assessment of the Glycemic Responses to Nutritional Products
Acronym: GLIN4
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nutricia Research (Industry)
Collaborators: INQUIS Clinical Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 24REX0080350
Record Dates: First submitted 2025-01-21; First posted 2025-01-28 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Glycemic Response
Keywords: Glycemic response; Glycemic Index; Nutritional products; Healthy Individuals

STUDY DESIGN:
Intervention Model Description: 10 products will be tested (7 test products and 3 controls)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (10):
- Arm 1 (Other): All subjects will receive all interventions during the trial. The order of the Nutritional products will be randomized.
  Interventions: Dietary Supplement: First Reference product
- Arm 2 (Other): All subjects will receive all interventions during the trial. The order of the Nutritional products will be randomized.
  Interventions: Dietary Supplement: Second reference product
- Arm 3 (Other): All subjects will receive all interventions during the trial. The order of the Nutritional products will be randomized.
  Interventions: Dietary Supplement: Third reference product
- Arm 4 (Other): All subjects will receive all interventions during the trial. The order of the Nutritional products will be randomized.
  Interventions: Dietary Supplement: First Concept product
- Arm 5 (Other): All subjects will receive all interventions during the trial. The order of the Nutritional products will be randomized.
  Interventions: Dietary Supplement: Second Concept product
- Arm 6 (Other): All subjects will receive all interventions during the trial. The order of the Nutritional products will be randomized.
  Interventions: Dietary Supplement: Third Concept product
- Arm 7 (Other): All subjects will receive all interventions during the trial. The order of the Nutritional products will be randomized.
  Interventions: Dietary Supplement: Fourth Concept product
- Arm 8 (Other): All subjects will receive all interventions during the trial. The order of the Nutritional products will be randomized.
  Interventions: Dietary Supplement: Fifth Concept product
- Arm 9 (Other): All subjects will receive all interventions during the trial. The order of the Nutritional products will be randomized.
  Interventions: Dietary Supplement: Sixth Concept product
- Arm 10 (Other): All subjects will receive all interventions during the trial. The order of the Nutritional products will be randomized.
  Interventions: Dietary Supplement: Seventh Concept product

INTERVENTIONS:
Dietary Supplement: First Reference product — dextrose (containing 25 grams of carbohydrates)
  Arms: Arm 1
Dietary Supplement: Second reference product — dextrose (containing 25 grams of carbohydrates)
  Arms: Arm 2
Dietary Supplement: Third reference product — dextrose (containing 25 grams of carbohydrates)
  Arms: Arm 3
Dietary Supplement: First Concept product — Plant-Based Oat Beverage with Sugar 1 (containing 25 grams of carbohydrates)
  Arms: Arm 4
Dietary Supplement: Second Concept product — Plant-Based Oat Beverage with Sugar 2 (containing 25 grams of carbohydrates)
  Arms: Arm 5
Dietary Supplement: Third Concept product — Plant-Based Oat Beverage with Sugar 3 (containing 25 grams of carbohydrates)
  Arms: Arm 6
Dietary Supplement: Fourth Concept product — Plant-Based Oat Beverage with Sugar 4 (containing 25 grams of carbohydrates)
  Arms: Arm 7
Dietary Supplement: Fifth Concept product — Plant-Based Oat Beverage No Sugar 1(containing 25 grams of carbohydrates
  Arms: Arm 8
Dietary Supplement: Sixth Concept product — Plant-Based Oat Beverage No Sugar 2 (containing 25 grams of carbohydrates
  Arms: Arm 9
Dietary Supplement: Seventh Concept product — High calorie, high protein oral powder nutritional supplement. (containing 25 grams of carbohydrates
  Arms: Arm 10

SUMMARY:
This study assesses the glycemic responses to nutritional products. During a study visit fasted subjects will consume one serving of the reference product or the test product. Capillary blood samples will be taken at baseline and at several time-points over a 2-hr period. Several nutritional products will be tested over time.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 and ≤ 65 years
2. Body mass index (BMI) between 18.5 and 27 kg/m²

Exclusion Criteria:

1. Baseline fasting Glucose ≥6.1 at screening visit
2. Known history of gastrointestinal disease, bariatric surgery, AIDS, hepatitis, a history or presence of clinically important endocrine (including Type 1 or Type 2 diabetes mellitus), or any condition which might, in the opinion of the medical director either: 1) make participation dangerous to the subject or to others, or 2)affect the results.
3. Use of medications known to influence carbohydrate metabolism, gastrointestinal function or appetite, including, but not limited to adrenergic blockers, diuretics, thiazolidinediones, metformin and systemic corticosteroids within 4 weeks of the screening visit, or any medication which might, in the opinion of the medical director either: 1) make participation dangerous to the subject or to others, or 2) affect the results.
4. Major trauma or surgical event within 3 months of screening.
5. Known intolerance, sensitivity or allergy to test products.
6. Extreme dietary habits, as judged by the Investigator (i.e. Atkins diet, very high protein diets, etc.).
7. History of cancer in the prior two years, except for non-melanoma skin cancer.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2025-01-23 (Actual); Primary Completion 2025-03-04 (Actual); Study Completion 2025-03-04 (Actual)

PRIMARY OUTCOMES:
The glycemic index of nutritional products | from enrollment to the end of treatment at about 9 weeks

SECONDARY OUTCOMES:
1. The postprandial glucose levels at each time point after each test product compared with the mean of the 3 references | from enrollment to the end of treatment at about 9 weeks
2. The postprandial incremental area under the curve (iAUC) after each test product compared with the mean of the 3 references | from enrollment to the end of treatment at about 9 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- INQUIS Clinical Research, Ltd , 20 Victoria Street, 3rd Floor, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No